CLINICAL TRIAL: NCT04889144
Title: Latinos' Beliefs and Communication About Advance Care Planning
Brief Title: PLAN Intervention to Enhance Engagement of Latino Cancer Patients in Advanced Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Megan Shen, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1121949; K07CA207580 (NIH); NCI-2022-00542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10760 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm
Keywords: advance care planning; Latinos; communication
MeSH Terms: conditions — Neoplasm Metastasis; Communication | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (PLAN intervention) (Experimental): Patients participate in PLAN intervention, consisting of 3 coaching sessions over 45-60 minutes each with a health coach.
  Interventions: Other: Communication Intervention; Other: Questionnaire Administration
- Arm II (Best practice) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Participate in PLAN intervention
  Arms: Arm I (PLAN intervention)
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (Best practice)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial tests whether Planning for Your Advance Care Needs (PLAN) intervention works to enhance Latino patients' understanding of and engagement in advanced care planning. The PLAN intervention may be an effective method to help people with cancer plan for and talk about advance care planning (the care they would want if they were unable to communicate) with their loved ones and doctors.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in PLAN intervention, consisting of 3 coaching sessions over 45-60 minutes each with a health coach.

ARM II: Patients receive usual care.

After completion of study treatment, patients are followed up at 1 week and then at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Identifying ethnically as Latino.
* Locally advanced or metastatic cancer and/or have experienced disease progression on at least first-line chemotherapy.
* Ability to provide informed consent.

Exclusion Criteria:

* Not fluent in English or Spanish.
* Severely cognitively impaired (as measured by Short Portable Mental Status Questionnaire scores of >= 6 to be delivered by trained study research staff during screening).
* Too ill or weak to complete the interviews (as judged by interviewer).
* Currently receiving palliative care/hospice at the time of enrollment (to allow prediction of [advanced care planning] ACP).
* Children and young adults under age 18.
* Patients deemed inappropriate for the study by their treating oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Shen, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - Weill Cornell Medicine, New York, New York
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Confluence Health, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that a total of n=27 patients enrolled in this study, n=22 completed baseline, and n=20 were randomized. As such, we can only provide baseline characteristics by intervention group for n=20 patients. Additionally, n=11 patients completed follow-up surveys, so all data reporting requiring follow-up data is provided for those n=11 patients.
Period: Overall Study
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Started | 11 | 9
Completed | 4 | 7
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Population: A total of n=27 patients enrolled in this study, n=22 completed baseline, n=20 were randomized (individuals we have data on baseline characteristics and arm/condition assignment), and n=11 we have baseline and follow-up data for. As such, baseline characeteristics are reported for n=20 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice) | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: For age, n=1 patient in the control condition did not provide a value so only n=8 are reported out of the n=9 who completed the baseline. Similarly, n=19 are reported out of n=20 for the overall column.
  years
    number analyzed (Participants) | 11 | 8 | 19
    (all) | 52.3 (9.31) | 50.2 (12.10) | 51.4 (10.29)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 8 | 4 | 12
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Please note, that we had a category for "Other (Hispanic/Latino)" as many patients do not identify with a racial category who identify as Hispanic/Latino. In this study, n=3 (intervention) and n=8 (control) who are listed as "Not reported" chose "Other (Hispanic/Latino)."
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 4 | 1 | 5
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Number/Proportion of Participants Who Completed the Intervention)
Description: Will be measured by intervention completion (Benchmark: >= 70% complete the intervention sessions).
Time Frame: Five weeks post-randomization (for intervention arm only)
Population: Please note: Only participants assigned to the intervention arm (Arm 1) were assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 11 | 0
Participants | 5 |

2. Primary Outcome: Acceptability (Helpfulness of the Intervention)
Description: Will be measured by a single-item question assessing helpfulness of the intervention (1 = not at all helpful, 5 = very helpful) as well an open-ended question about helpfulness of the intervention ("What was helpful about the intervention?") (Benchmark: >= 70% rate it as "helpful" or "very helpful"). Data reported as a count number of those who reported "4=helpful" or "5=very helpful" to this question.
Time Frame: Five weeks post-randomization (for intervention arm only)
Population: Please note: Only participants who completed the intervention were assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 5 | 0
Participants
  Reported "4=helpful" | 0 |
  Reported "5=very helpful" | 5 |

3. Primary Outcome: Change in Knowledge of Advance Care Planning
Description: Knowledge subscale of the Advance Care Planning Engagement survey, which is a 49-item scale with high reliability (Cronbach's alpha = .94). Subscale is 6 items with Likert-type answers ranging from 1=not at all to 5=extremely. Responses to these 6 items are summed to create total scores, ranging from 6 (low levels of knowledge) to 30 (high levels of knowledge). Higher scores indicate higher levels of knowledge. Mean score differences were calculated between baseline and follow-up for each study arm and tested for significance.
Time Frame: Baseline, five weeks post-randomization (after randomizing and completing the 3-week intervention if assigned)
Population: Due to the small sample size, inferential statistics were not run. Only participants who completed all study activities (e.g., follow-up surveys) were assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 4 | 7
score on a scale | 2.75 (3.40) | 1.86 (3.48)

4. Primary Outcome: Change in Readiness/Motivation to Engage in Advance Care Planning
Description: Readiness/motivation subscale of the Advance Care Planning Engagement survey, which is a 49-item scale with high reliability (Cronbach's alpha = .94). Subscale is 10 items with Likert-type answers ranging from 1=not at all to 5=extremely. Scores from these items are summed to created total scores, ranging from 10 (low level of readiness/motivation) to 60 (high level of readiness/motivation). Higher scores indicate higher levels of readiness/motivation. Mean score differences were calculated between baseline and follow-up for each study arm and tested for significance.
Time Frame: Baseline, five weeks post-randomization (after randomizing and completing the 3-week intervention if assigned)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 4 | 7
score on a scale | 10.0 (18.89) | 1.0 (6.08)

5. Primary Outcome: Change in Self-efficacy to Engage in Advance Care Planning
Description: Self-efficacy subscale of the Advance Care Planning Engagement survey, which is a 49-item scale with high reliability (Cronbach's alpha = .94). Subscale is 6 items with Likert-type answers ranging from 1=not at all to 5=extremely. These items are summed to create total scores, ranging from 6 (low levels of self-efficacy) to 30 (high levels of self-efficacy). Higher scores indicated higher levels of self-efficacy. Mean score differences were calculated between baseline and follow-up for each study arm and tested for significance.
  Data reported is the mean change in this outcome from pre-randomization/baseline to post-randomization.
Time Frame: Baseline, five weeks post-randomization (after randomizing and completing the 3-week intervention if assigned)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 4 | 7
score on a scale | 0.00 (4.27) | 0.86 (5.30)

6. Primary Outcome: Change in Engagement in Advance Care Planning (End-of-life Care Discussions)
Description: End-of-life care discussions will be measured by asking patients to self-report whether they have discussed any of the following: (1) wishes they have about the care they would like to receive if they were dying and/or (2) advance care directives, with an oncology provider or family member: DNR orders, living wills, durable powers of attorney for health care (yes/no format). Engagement will be measured as a count to the degree to which they engaged in each of these, with no=0 and yes=1. Total score can range from 0 (low or none) to 8 (high or discussed all domains with providers and family). Data reported is the mean change in this outcome from pre-randomization/baseline to post-randomization,
Time Frame: Baseline, five weeks post-randomization (after randomizing and completing the 3-week intervention if assigned)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 4 | 7
score on a scale | 2.50 (1.73) | 1.29 (3.20)

7. Primary Outcome: Change in Completion of Advance Directives
Description: Completion of advance directives will be assessed by examining the medical chart for completed advance directive documents (DNR order, living will, health care proxy/durable power of attorney). Completion will be measured as a count to the degree to which they completed each of these, with no=0 and yes=1. Scores can range from 0 (low or none completed) to 3 (high or all completed). Data reported is the mean change in this outcome from pre-randomization/baseline to post-randomization.
Time Frame: Baseline, five weeks post-randomization (after randomizing and completing the 3-week intervention if assigned)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
Number analyzed (Participants) | 4 | 7
score on a scale | 0.0 (0.82) | 0.43 (0.53)

ADVERSE EVENTS:
Time Frame: All participants were monitored for AEs/SAEs during the entire enrollment period from the point of consent until the final follow-up survey. This time frame was up to n=11.6 weeks (maximum) and was n=4.0 weeks on average.
Description: We did both systematic reporting (checking medical records for hospitalizations and/or death) as well as non-systematic reporting (noting when a patient mentioned distress, hospitalization, etc.).
Arm/Group | Arm I (PLAN Intervention) | Arm II (Best Practice)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT04889144/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT04889144/ICF_000.pdf